CLINICAL TRIAL: NCT04066153
Title: Patient Reported Unmet Needs for Function and Supportive Occupational- and Physiotherapy Rehabilitation Interventions in a Palliative Care Setting
Brief Title: Patient Reported Unmet Needs for Function and Supportive Occupational- and Physiotherapy Rehabilitation Interventions
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jan Christensen, post doc, Rigshospitalet, Denmark
Other Study IDs: 2018-418 6670
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Kidney Diseases; Heart Failure; Neurologic Disorder; Liver Diseases; Pulmonary Disease; Side Effect; Quality of Life; Physical Disorder
Keywords: Palliative care; Physical functioning; Unmet needs
MeSH Terms: conditions — Neoplasms; Kidney Diseases; Heart Failure; Nervous System Diseases; Liver Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Purpose: To determine unmet functional needs in patients referred to the Palliative Care Unit at Rigshospitalet, Copenhagen University Hospital will be asked to fill out self reported questionnaires regarding problem intensity, problem burden and felt needs, physical functioning, emotional functioning, fatigue, sleep, distress. Furthermore patients physical function will be evaluated.

DETAILED DESCRIPTION:
Physical functioning is found to be an important predictor for survival and physical ability 'to do what one wants' affects quality of life in cancer patients in palliative care and their spouses. Despite this, physical functioning is reported as a neglected dimension in palliative care quality of life outcome measures, and advanced cancer patients report that they do not receive the help they need. The vast majority of patients with advanced cancer described unmet palliative care needs, and with the most frequently reported problems being; fatigue (73%), limitations doing physical activities (65%), limitations in work and daily activities (58%), worry (58%), difficulties with sexuality (54%), pain (52%) and problems with concentration (43%). Furthermore, limitations in physical functioning and physical activity is a leading cause of distress and psychological problems a rehabilitative approach in palliative care integrated in the interdisciplinary interventions to the patients must be maintained throughout the entire illness trajectory from diagnosis through treatment, rehabilitation and palliative care to address such problems.

However, prevalence of patient unmet needs and reported physical functioning and performance is reported to differentiate largely between palliative units.

In order to address the functional needs of patients receiving specialist palliative care studies of their specific needs are required. Therefore, the aim of this study is to investigate the patient reported unmet needs for function and supportive occupational- and physiotherapy rehabilitation interventions in the palliative unit at Copenhagen University Hospital, Rigshospitalet. Furthermore, we aim to investigate if observations, additional disease-specific patient reported outcomes and assessment of physical function and performance can support the unmet needs.

ELIGIBILITY:
Inclusion Criteria :

All adult patients (≥ 18 years) referred to the Palliative Care Unit at Copenhagen University Hospital, Rigshospitalet.

Exclusion Criteria:

Inability to read and understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥ 18 years) referred to the Palliative Care Unit at Copenhagen University Hospital, Rigshospitalet will be considered eligible for inclusion. Patients will be cancer and non-cancer patients, some will receive in-hospital treatment at the hospital and others outpatient treatment.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Unmet physical functioning needs | At baseline
  The Three-Levels-of-Needs Questionnaire (3LNQ)

SECONDARY OUTCOMES:
Lower body physical function | At baseline
  30 seconds Sit-To-Stand test
Hand grip strength | At baseline
  Maximum strength test by handgrip dynamometer
Walking endurance | At baseline
  Six Minute Walking Test
Health-related quality of life | At baseline
  EORTC QLQ-C30
Overall distress | At baseline
  Distress thermometer
Psychological distress | At baseline
  Hospital Anxiety and Depression Scale (HADS)
Sleep quality | At beseline
  Pittsburgh Sleep Quality Index (PSQI)
Level of fatigue | At baseline
  Functional Assessment of Cancer Therapy - Fatigue (FACT-F) 13 item fatigue subscale
Patients self-perception of performance in everyday living | At baseline
  The Canadian Occupational Performance Measure (COPM)
Physical activity level | At baseline
  International Physical Activity Questionnaire (IPAQ) short form

CONTACTS AND LOCATIONS:
Overall Officials: Jan Christensen, Principal Investigator — Department of Occupational- and Physiotherapy, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32788277/